CLINICAL TRIAL: NCT03687528
Title: Platelet Inhibitor Treated Patients With Head Injury Trauma Without Any Clinical Symptoms of Cerebral Haemorrhage (NICE Criteria) : is the CT-scan Mandatory ?
Brief Title: Platelet Inhibitor Treated Patients With Head Injury Trauma Meeting NICE Criteria : is the CT-scan Mandatory ?
Acronym: TCAP
Status: Recruiting | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC17_8839_T.CAP
Record Dates: First submitted 2018-09-26; First posted 2018-09-27 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Head Injury Trauma; Emergencies
Keywords: emergencies; platelet inhibitors; minor head injury trauma; CT-scan
MeSH Terms: conditions — Emergencies | interventions — Tomography Scanners, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with minor head injury trauma: The emergency protocol for antiplatelet inhibitors treated patient with head injury trauma and meeting others NICE criteria involves a clinical exam followed by a CT-scanner.
  Interventions: Radiation: CT-scanner

INTERVENTIONS:
Radiation: CT-scanner — After a clinical exam, patient have a CT-scanner to check any cerebral haemorrhage.

SUMMARY:
At the emergencies rooms, patients with head trauma meeting one of the NICE criteria, which include antiplatelet inhibitors treatment, are considered as patients with a risk of cerebral haemorrage and are taken systematically for a CT-scanner.

However, there are more and more antiplatelet inhibitor's patient with minor head injury traumas seen at the emergencies room and the efficiency of this NICE criteria is controversial on litterature.

This study aims to determine that the absence of no other NICE criteria than antiplatelet inhibitors is a sufficient condition to eliminate a cerebral haemorrhage for patients with head injury traumas, and conversely, that antiplatelet inhibitors treatment would not be by itself an indication for a CT-scanner.

DETAILED DESCRIPTION:
Head injuries are a frequent reason for emergency services, and according to studies, they represent between 5% and 10% of patients treated in emergencies. Among them, 90% are minor head injury traumas. NICE criteria has been defined to establish patients who need a CT-scanner because of a risk of cerebral haemorrhage.

NICE criteria include several conditions including taking antiplatelet inhibitors. However, the real risk of cerebral haemorrhage for theses cases is controversial in litterature. In parallel, more and more patients undergoing antiplatelet inhibitor's treatment are seen in emergencies after a head injury trauma.

In routine protocol at the emergency rooms, these patients are seen for a clinical exam and next submitted to a CT-scanner. If the clinician can't detect a cerebral haemorrage, the patient will return at home.

This study aims to determine that the absence of no other NICE criteria than antiplatelet inhibitors treatment is a sufficient condition to eliminate a cerebral haemorrhage for patients with head injury traumas, and conversely, that antiplatelet inhibitors treatment would not be by itself an indication for a CT-scanner.

This is a diagnostic, case-only, prospective, multicenter study with a blinded primary outcome measure assessment.

As described in routine protocol, in this study antiplatelet inhibitor's patients with head injury trauma will be seen for a clinical exam and next submitted to a CT-scanner. After a month, patient will be called by the clinical center to ask about morbidity and mortality. Especially, clinicans will report on the emergence of a cerebral haemorrhage during this month.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Patient with a head injury trauma, described by the patient or seen at the clinical exam
* Glasgow score between 13 and 15 at the clinical exam
* Current treatment with antiplatelet inhibitors
* Informed non opposition form signed

Exclusion Criteria :

* Absence of CT-scanner
* Patients with double anti-platelet aggregation
* Patients on anticoagulants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major patients undergoing antiplatelet inhibitors treatment which are reported at the clinical exam as having a head injury trauma.
  These patients don't meet another NICE criteria :
  * neurological focal deficit
  * amnesia for more than 30 min
  * glasgow score less than 15 after 2 hours
  * loss of consciousness associated with either a high velocity or an age > 65 years old
  * suspicion of a cranial open fracture
  * fracture on cranial basis
  * more than 1 vomit
  * post-traumatic convulsion
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Existence of a cerebral haemorrhage at the CT-scanner. | 1 day
  Cerebral haemorrhage seen at the CT-scanner.

SECONDARY OUTCOMES:
Neurosurgeries' rate after one month | 1 month
  Neurosurgeries' rate after one month
Existence of a cerebral haemorrhage associated to death | 1 month
  Existence of a cerebral haemorrhage associated to death
Existence of a cerebral haemorrhage associated to neurosurgery | 1 month
  Existence of a cerebral haemorrhage associated to neurosurgery
Existence of a cerebral haemorrhage associated to hospitalization with more than 24h of intubation | 1 month
  Existence of a cerebral haemorrhage associated to hospitalization with more than 24h of intubation
Existence of a cerebral haemorrhage associated to more than 2 nights at hospital | 1 month
  Existence of a cerebral haemorrhage associated to more than 2 nights at hospital
Death rate after one month | 1 month
  Death rate after one month

CONTACTS AND LOCATIONS:
Overall Officials: Paul-Georges REUTER, Pr, Study Director — CHU Rennes
Locations (12):
- France (12):
  - CHU d'Angers, Angers
  - CHU Brest, Brest
  - CH Chartres, Chartres
  - CH Le Mans, Le Mans
  - CH Bretagne Sud, Lorient, Lorient
  - CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - CH Bretagne Sud - Quimperlé, Quimperlé
  - CHU de Rennes, Rennes
  - CH de Saint Brieuc, Saint-Brieuc
  - CH de Saint Malo, St-Malo
  - CH Bretagne Atlantique, Vannes

IPD SHARING:
Plan to Share IPD: Undecided